CLINICAL TRIAL: NCT02807220
Title: A Phase 4, Single Arm Trial Assessing the Efficacy and Safety of Imuneks 10 mg Capsules in the Prophylaxis of Cold and the Maintenance of the Good Health State in Healthy Subjects
Brief Title: Efficacy and Safety of Imuneks 10 mg Capsules in the Prophylaxis of Cold
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imuneks Farma ilac San. Tic. A.S. (Industry)
Collaborators: TC Erciyes University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ALPAN-KA001-16
Record Dates: First submitted 2016-06-08; First posted 2016-06-21 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Cold Symptoms
Keywords: Imuneks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imuneks 10mg (Experimental): Two capsules of the study drug every morning approximately two hours after breakfast for six weeks
  Interventions: Drug: Imuneks 10mg

INTERVENTIONS:
Drug: Imuneks 10mg — Two capsules of the study drug every morning approximately two hours after breakfast for six weeks
  Other Names: micronized Beta-1,3/1,6-D-glucan

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of Imuneks 10 mg Capsules in the prophylaxis of cold and the maintenance of the good health state in 70 healthy subjects.

DETAILED DESCRIPTION:
Study Design: A Phase 4, single arm, efficacy and safety study.

Phase: Phase IV

Number of Sites: 1 (one)

Study Population: 70 healthy subjects of both genders. (This study is designed as a Phase 4 study aiming to obtain efficacy and safety data from the study group. Estimation of Sample Size and Power for Comparing Two Means with standard deviation for each primary endpoint was performed for determination of the study population. 70 healthy subjects were estimated to be sufficient for obtaining efficacy and safety data from the study group.)

Study Drug: Imuneks 10 mg Capsules, containing 10 mg micronized Beta-1,3/1,6-D-glucan derived from baker's yeast of which at least 80 % is below 10 microns (İMUNEKS FARMA İlaç Sanayi ve Ticaret A.Ş., Turkey)

Procedure: Subjects will receive two capsules of the study drug every morning approximately two hours after breakfast

Patients Registry: Study staff will maintain appropriate medical and research records for this study, in compliance with ICH E6 and regulatory and institutional requirements for the protection of confidentiality of subjects. Study staff will permit authorized representatives of regulatory agencies to examine (and when required by applicable law, to copy) research records for the purposes of quality assurance reviews, audits, and evaluation of the study safety, progress and data validity.

The results from screening and data collected during the study will be recorded in the subject's Case Report Form.

MedDRA Data dictionary will be used for adverse event determination and normal laboratory ranges will be added to the ITF.

Standardized CRFs will be used to document the subjects' data during the course of the study. The investigator will assure that all data are entered promptly, legibly, completely, accurately and in accordance with source documents. This also applies to the data for those subjects who -after having consented to participate -underwent baseline examinations required especially for inclusion into the study but who - because a criterion for exclusion was met or for other reasons - were not included into the study.

The Sponsor will require the top (original) copy of the CRF but the Investigator will also be left with a copy for his trial file.

Each page of the CRF must be signed by the (co-)Investigator. A stamp as signature is not allowed.

Any corrections to the case report forms must be carried out by the investigator or his designate. A single line must be drawn through the original entry, making sure the previous data are not totally obliterated. The reason for the correction has to be given and it has to be dated and initialled. Incorrect entries must not be covered with correcting fluid, or obliterated, or made illegible in any way.

Even if there are no changes from a previous examination, in the interests of completeness of data acquisition, the questions which are repeated in each section of the case report forms should be answered in full text. A reasonable explanation must be given by the investigator for all missing data.

The case report forms will be completed immediately after termination of the individual treatment and observation periods and the final examination. After being signed by the Principal Investigator, they will be sent to QC department for data verification. Thereafter, CRFs will corrected, if applicable. CRFs cannot be sent by post but only be personally submitted to the monitor during a visit.

All medical records upon which the case report forms are based must be kept for at least 5 years after completion of the study. At this time it will be discussed with the Sponsor whether or not storage is required for a longer period. It is the responsibility of the investigator to assure that the study is conducted in accordance with the protocol and that valid data are entered into the CRF.

Monitoring and auditing of this study will be conducted in accordance with SOPs (IDEAL-BE-S08-1, IDEAL-BE-S08-2 and IDEAL-BE-S08-3) developed by IDEAL in order to check the adherence to the protocol in compliance with Good Clinical Practice guidelines and to ensure international acceptability of the study data. In support of these measures, the investigator will make the records available to ALPAN, IDEAL or to the Sponsor upon request at reasonable times. Case report forms will be checked for completeness and clarity.

Data verification is legally required and will be done by direct comparison with source documents in case of subject's respective consent or by cross-checking with source documents in the presence of the investigator - always giving due consideration to data protection and medical confidentiality. In this respect the investigator assures ALPAN and IDEAL of support at all times.

The investigator will permit a representative of ALPAN, IDEAL or the Sponsor to monitor the study as frequently as necessary to determine that data recording and protocol adherence are satisfactory. The CRFs and related documents will be reviewed in detail in accordance with the SOPs of IDEAL(IDEAL-BE-S08-1, IDEAL-BE-S08-2 and IDEAL-BE-S08-3) and Good Clinical Practice regulations.

Visits may be conducted also by a representative of ALPAN, IDEAL or the Sponsor at suitable intervals throughout the study. These visits will be for the purpose of verifying adherence to the protocol and the completeness and exactness of the data entered on the Case Report Forms. The Sponsor is allowed to get any information about the state of the study. Case Report Forms will be transported from the investigator via IDEAL to the Sponsor after completion of the trial.

In fulfilment of their obligation to the Sponsor to verify compliance with the protocol, ALPAN and IDEAL will require that the investigator permits their monitors to review those portions of the subject's primary medical records which directly concern this study.

It is the investigator's obligation to assure documentation of all relevant data in the subject's file, such as medical history / concomitant diseases, date of study enrolment, visit dates, results of examinations, administrations of medication and adverse events.

The investigator will affirm and uphold the principle of the subject's right for protection against the invasion of privacy. Throughout the study, all data will only be identified by volunteer number. The data will be blinded correspondingly in all data analyses.

In order to guarantee that the performance of the study is in accordance with the GCP provisions, in-house and, if needed, on-site audits may be carried out. The auditor will be independent from the staff involved in the proceedings of this clinical study.

The investigator agrees to give the auditor access to all relevant documents for review. The same applies in case of an inspection of local or national authorities.

After every on-site audit the investigator will receive an audit confirmation by the auditor. This has to be filed together with the study documentation and be made available to the local authorities in case of supervision. At the end of the study, an audit certificate will be included in the final report.

Safety Monitoring: Adverse event questioning and examination will be done at every visit.

Evaluation Criteria:

Primary Endpoints:

* Difference from baseline of Imuneks 10 mg Capsules on the immunological examinations (lymphocytes, macrophages, neutrophils, eosinophils and monocytes)
* Proportion of subjects with no symptoms of cold(colds seen in the first week will be excluded from the evaluations as prophylactic effect will not be assessable before this period)

Secondary Endpoint:

• Number of Subjects Reporting Side Effects and number of subjects who took rest periods during the treatment period.

Plan for missing data:

Subjects who prematurely withdraw from treatment or from the trial will not be replaced. Missing values for all efficacy parameters will not be included to the evaluation. Missing values will be treated using a list wise deletion method.

All computations will be performed by commercial statistical software such as SPSS®, SAS® or WinNonlin®. Microsoft Excel may be used for tabulation of the data and description statistics. Graphical summaries will be presented in SAS® or WinNonlin® format.

A detailed description of the analyses to be performed will be provided in the statistical analysis plan.

Statistical Considerations: Populations for Analysis: Intent-to Treat (ITT) population will be primary analysis population. Per Protocol (PP) Population will be supportive analysis population for analysis.

The descriptive statistics: Arithmetic mean (MEAN), standard deviation (SD), coefficient of variation (%CV), maximal value (MAX), minimal value (MIN), and median value (MEDIAN) will be applied for applicable demographic and immunological data and presented in tables.

Efficacy Analysis: Primary Endpoints will be evaluated by either paired t-tests or Wilcoxon signed-rank test for two-group comparisons. Repeated measures ANOVA or Friedman test will be applied for more than two-group comparisons. All p values will be two-tailed; p< 0.05 denoted statistical significance.

Planned Initiation: October 2016 (inclusion of first subject)

Study Duration: 1 month for enrolment + 6 weeks follow-up and evaluation

Sponsor: İMUNEKS FARMA İlaç Sanayi ve Ticaret A.Ş. Prof. Dr. Bülent Tarcan Cad. Pak İş Merkezi No:5 Gayrettepe-Beşiktaş/İstanbul Representatives: Mehmet Nevzat Pisak and Dr. Gökhan Demir Version Number: Draft 2.0 Version Date: 16 May 2016

o Standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management.

ELIGIBILITY:
Inclusion Criteria:

* physically and mentally healthy as judged by means of a medical and laboratory standard
* the outcome of the following examinations should be clinically insignificant: medical and surgical history (hypo-, hypertension, allergy, other diseases, major surgery, micturition, defecation, sleep, illness within the last 4 weeks prior to the start of the trial)
* life style and habits (consumption of alcohol, nicotine, coffee, tea, coke, special diet, drug abuse) should be normal/acceptable
* body temperature, pulse rate, blood pressure, 12 lead ECG should be normal/acceptable.
* physical examination (general state and abnormal findings per system: endocrine/metabolic, allergies, drug sensitivities, head, neck, eyes, ears, nose, throat, cardiovascular, respiratory, gastrointestinal, hepatic/biliary, urogenital, musculoskeletal, Iymph nodes, skin, and neurological/psychiatric) should be normal/acceptable
* laboratory examination (blood/serum examination: sodium, potassium, calcium, chloride, total protein, glucose, creatinine, BUN, uric acid, total bilirubin, AST, ALT, GGT, ALP, haemoglobin, haematocrit, erythrocytes, Ieukocytes, platelet count; HBsAg, HIV-Ab, HCV-Ab; urine examination: urine pH, protein, glucose, ketones, blood, Ieukocytes, bilirubin, nitrites and sediment) should be normal/acceptable.
* normal body weight in relation to height and age according to weight(kg) BMI = (accepted range 18.5 and30 kg/m2) height (m)2
* subjects must be competent to sign and have signed a consent form before study entry

Exclusion Criteria:

* acute or chronic upper airways disease, chronic cough, chronic rhinitis (e.g. allergic rhinitis) or asthma,
* vaccination against influenza or swine flu
* within 21 days before the study start, suspected swine flu or influenza, body temperature 38 0C,
* pregnancy or nursing,
* use of immunosuppressant, stimulants or common cold therapeutics,
* bacterial tonsillitis,
* allergic diathesis or any clinically significant allergic disease (i.e. asthma)
* any history of drug hypersensitivity (especially to β-glucan and related compounds)
* presence or a history of clinically significant cardiovascular, renal, hepatic, pulmonary, metabolic, endocrine, haematological, gastrointestinal, neurological, psychiatric or other major diseases
* clinically significant illness within 4 weeks before the start of the study
* intake or administration of any prescribed systemic or topical medication within 2 weeks prior to the start of the study; in the case of intake or administration of any prescribed systemic or topical medication within 4 weeks before the start of the study because of an insignificant illness, this should be stated in the CRF.
* intake or administration of OTC medication (including herbal remedies) within 1 week prior to the start of the study
* concomitant intake or administration of any systemic or topical drugs (including herbal remedies)
* treatment with any investigational drug (i.e., drug not yet approved) in the last 2 months (60 days) before beginning of the trial
* medication with drugs known to alter organs or systems such as barbiturates, phenothiazines, cimetidine, omeprazole etc. within the last 2 months (60 days)
* major surgery of the gastrointestinal tract except for appendectomy
* supine blood pressure, after resting for 5 min, higher than 140/90 or lower than 100/60 mmHg
* supine pulse rate, after resting for 5 min, outside the range of 50 - 90 beats/min
* any clinically significant abnormality of the ECG (12 leads) recorded in rest
* laboratory values outside the normal range (Appendix 5) with clinical relevance at entry examination
* alcohol abuse i.e. regular use of more than 2 units of alcohol per day or a history of alcoholism or drug/chemical abuse (one unit of alcohol equals ½ l of beer, 200 ml wine or 50 ml of spirits) or recovered alcoholics
* vegetarian or any special diet due to any reason
* knowledge to have any type of parenterally transmitted hepatitis or carrier of the HBsAg (HBsAg test positive)
* HIV-Ab test positive
* Test on anti-HCV antibodies positive
* legal incapacity and/or other circumstances rendering the subject unable to understand the nature, scope and possible consequences of the study
* evidence of an uncooperative attitude
* > 10 % non-compliance to the investigational product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

PRIMARY OUTCOMES:
Prophylaxis of common cold and the change in blood lymphocyte, macrophage, neutrophil, eosinophil and monocyte counts from baseline values after first, third and sixth weeks after the oral use of the study medication. | 6 weeks
  The baseline will be established by taking blood samples from the participants at their first visits.
  Each participant will report to the study staff any symptoms such as runny nose, cough, nasal congestion and sneezing during 6 weeks after administering the first dose of the study medication. Cold symptoms seen in the first week will be excluded from the evaluations as prophylactic effect will not be assessable before this period.

SECONDARY OUTCOMES:
The number of participants who took sick leaves. | 6 weeks
  The participants who will take sick leaves form their work during the study will be reported.
Number of Participants with Adverse Events That Are Related to The Study Medication. | 6 weeks
  The number of Participants with Adverse Events that are related to the study medication during the study period will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet İnal, Asst. Prof., Principal Investigator — Erciyes University Hakan Çetinsaya İKU Merkezi (Center for GCP)
Locations (1):
- Erciyes University Hakan Çetinsaya İKU, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
According to Turkish laws it is forbidden to share personal data